CLINICAL TRIAL: NCT04241380
Title: Anticoagulation Medicine in Surgical Repair for Total Anomalous Pulmonary Venous Connection: a Randomize Multi-centers Study
Brief Title: Anticoagulation Medicine in Surgical Repair for Total Anomalous Pulmonary Venous Connection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019050505
Record Dates: First submitted 2020-01-17; First posted 2020-01-27 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-01

CONDITIONS: Total Anomalous Pulmonary Venous Connection
Keywords: Total anomalous pulmonary venous connection (TAPVC); Anticoagulant management; Pulmonary venous obstruction (PVO); outcomes
MeSH Terms: conditions — Scimitar Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional treatment group (Active Comparator): Patients in this group will received conventional treatments. Drug: None. Drug: For the high-risk patients, doctors will assess their risk factors and choose continuous infusion heparin (initial dose 10 iu/kg/h and dynamic regulation until the activated coagulation time (ACT) 160-180 s) if needed. Aspirin 5 mg/kg may be given every eight hours subsequently for 3 months.
  Interventions: Other: No anticoagulant solutions; Drug: Anticoagulant management
- Anti-coagulant treatment (Experimental): Continuous infusion heparin. Patients in this group will received continuous infusion heparin 6 hours postoperatively (initial dose 10 iu/kg/h, dynamic regulation according to ACT 160-180s). After the removal of deep vein catheter, aspirin 5mg/kg will be given every eight hours subsequently for three months. Study will follow the intention-to-treat principle.
  Interventions: Drug: Anticoagulant Solutions

INTERVENTIONS:
Drug: Anticoagulant Solutions — Patients in this group will received continuous infusion heparin 6 hours postoperatively (initial dose 10 iu/kg/h, dynamic regulation according to ACT 160-180s). After the removal of deep vein catheter, aspirin 5 mg/kg will be given every eight hours subsequently for 3 months.
  Other Names: Continuous infusion heparin
  Arms: Anti-coagulant treatment
Other: No anticoagulant solutions — They will receive non-coagulant or coagulant treatment according to clinical conditions.
  Arms: Conventional treatment group
Drug: Anticoagulant management — Continuous infusion heparin (initial dose 10 iu/kg/h and dynamic regulation until the activated coagulation time (ACT) 160-180 s) for a few days.
  Aspirin 5 mg/kg will be given every eight hours subsequently for 3 months.
  Arms: Conventional treatment group

SUMMARY:
Total anomalous pulmonary venous connection (TAPVC) is a complex congenital heart disease, requiring surgical repair. Pulmonary venous obstruction (PVO) is the major complication, with limited effective reinterventions and poor outcomes. This trial aims at investigating that postoperative anticoagulant management reduce the incidence of PVO.

DETAILED DESCRIPTION:
Total anomalous pulmonary venous connection (TAPVC) is a complex congenital heart disease, with all the pulmonary veins connecting to the right heart system through collateral vessels, accounts for about 3% of congenital heart disease. Pulmonary venous obstruction (PVO) is a major complication, with limited effective reinterventions and poor outcomes. The major challenge for surgical repair of TAPVC is to lower the incidence of PVO.

Previous studies in our center showed the abnormal coagulation function, such as elevated International Normalized Ratio (INR), and decreasing of prothrombin activity, are associated with a higher rate of PVO. Some researches suggested that postoperative application of anticoagulants might reduce the incidence of PVO, however, the evidences are still limited. This trial will randomize patients to receive either conventional postoperative management or continuous infusion anticoagulant (Heparin) until the removal of deep vein catheter. The primary endpoint will be incidence of PVO, days of chest drainage more than 40ml/d, and mortality rate. Secondary endpoints including readmission, functional capacity assessment, quality of life and incidence of complications will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* 1. Infants and neonates who are diagnosed with TAPVC
* 2. Infants and neonates who undergo initial surgical repair for TAPVC

Exclusion Criteria:

* 1. Concommitant diagnosis including functional single ventricular, double outlet right ventricle, tricuspid atresia, pulmonary atresia or transposition of the great arteries.
* 2. Older than 1-year-old.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2020-02-20 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative pulmonary venous obstruction (PVO) | 2 years
  The postoperative PVO were diagnosed by echocardiography or computed tomography scan
Days of chest drainage | 2 years
  > 40ml/d, assessed during inhospital stay
Mortality rate | 2 years
  Inhospital or during follow-up, exclude the discharge from hospital against doctors' suggestions.

SECONDARY OUTCOMES:
Level of coagulation indexes. | 2 years
  Blood samples were measured by coagulation function test during follow-up
Change in resting oxygen saturation | 2 years
  Answer question through telephone or other communication
Value of tricuspid annular plane systolic excursion | 2 years
  Measured by echocardiology from follow-up
Level of brain natriuretic peptide (BNP) | 2 years
  Measured during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhuang, M.D., Ph D., Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No